CLINICAL TRIAL: NCT03662867
Title: Application of Mindfulness Training in a Family-based Intervention for Improving Early Child Development and Stress Management in Economically Disadvantaged Families
Brief Title: Applying Mindfulness for Economically Disadvantaged Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21611415
Record Dates: First submitted 2017-09-20; First posted 2018-09-10 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2017-09

CONDITIONS: Stress
Keywords: mindfulness training; economically disadvantaged families; family-based interventions
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-based mindfulness intervention (Experimental): Family-based mindfulness intervention is a parallel-group intervention containing one parent program and one child program. The parent mindfulness program lasts for 6 weeks, one session per week, and each session lasts for 1.5 hours. The child mindfulness program lasts for 8 weeks, one session per week, and each session lasts for 1 hour. In the fourth and sixth sessions of the parent program, 30-minute joint practice of parents and children is incorporated. All sessions are implemented by qualified instructors.
  Interventions: Behavioral: Family-based mindfulness intervention
- Wait-list control (Other): Intervention group participants were assessed at baseline (T1) and after the intervention (T2). Control group participants were assessed at the same time with the intervention group, and would receive the same program after posttest of intervention groups.
  Interventions: Other: Wait-list

INTERVENTIONS:
Behavioral: Family-based mindfulness intervention — For the parent program of family-based mindfulness intervention, the content includes: guide body scan practice; guide stretching exercise and mindful breathing; guide practice of mindfulness to breath and body; teach three-minute breathing exercise; guide joint session and let parents practice mindfulness with children; guide mindfulness practice of exploring difficulties; and teach loving-kindness practice.
  For the child program, the content includes: guide mindful breathing exercise; guide mindful movement exercises; use stories of animal characters to guide body scan exercise; guide mindful eating and mindful walking exercise; tell stories about different emotions and guide discussion; guide the imagination exercise about different emotions; and guide loving-kindness practice.
  Arms: Family-based mindfulness intervention
Other: Wait-list — No intervention is given between T1 and T2. Family-based mindfulness intervention would be received after posttest of intervention groups.
  Arms: Wait-list control

SUMMARY:
The purpose of this study is to assess the effectiveness of a family-based mindfulness intervention (FBMI) in reducing parental stress and promoting child adjustment. Intervention effectiveness will be tested by conducting a randomized controlled trial comparing a group receiving FBMI to a wait-list control group. Children aged five and their parents will be recruited to participate in the study. Eligible families will be recruited, stratified by level of economically disadvantage, behaviour problem scores, and parental stress, and then randomly assigned to the two groups. Intervention groups will be conducted by instructors with professional training. Children in the intervention group are expected to show improvements in cognitive and language development, behaviour problems, attention and emotional/behavior regulation, and physiological stress (reduced cortisol and heart rate variability), compared with the waitlist control group. Parents are expected to show improvements in physiological and psychological stress, and mindfulness, compared with the waitlist control group.

DETAILED DESCRIPTION:
Economic disadvantage has been found to be associated with delayed cognitive and language development, and mental health symptoms such as aggression, anxiety of children. Chronic cumulative stressors of poverty disrupt their attention, emotional and behavioural regulation, that would further lead to negative impact in early development. As their parents are also affected by stress, they often become unresponsive, harsh and inconsistent in child discipline, resulting in a chronic stress to their children. Mindfulness is defined as paying attention purposefully and non-judgmentally to the present moment. It has been shown to improve attention, promote exposure to unpleasant experiences, facilitate cognitive change, and enhance the ability to cope with life stress. Mindfulness training has been established as an evidence-based intervention for people suffering from various chronic conditions. Its application in a family context, including parents and children, is just beginning. The purpose of this study is to assess the effectiveness of a family-based mindfulness intervention (FBMI) in reducing parental stress and promoting child adjustment. Intervention effectiveness will be tested by conducting a randomized controlled trial comparing a group receiving FBMI to a wait-list control group. Children aged five and their parents will be recruited to participate in the study. Eligible families will be recruited, stratified by level of economically disadvantage, behaviour problem scores, and parental stress, and then randomly assigned to the two groups. Intervention groups will be conducted by instructors with professional training. Children in the intervention group are expected to show improvements in cognitive and language development, behaviour problems, attention and emotional/behavior regulation, and physiological stress (reduced cortisol and heart rate variability), compared with the waitlist control group. Parents are expected to show improvements in physiological and psychological stress, and mindfulness, compared with the waitlist control group. The proposed project will be the first of its kind to use mindfulness training in a family context in Hong Kong. It is also unique as it examines the effectiveness of a mindfulness-based intervention with multiple outcome measures related to stress, combining self-reported measures with biomarkers, and psychological tests. For model building and theory development, this study may shed light on assessing the change mechanisms for promoting child learning, emotional and behavioural regulation, particularly in relation to studies of stress physiology and economically disadvantaged families. The results may not only benefit in Hong Kong but also those in other Chinese societies and countries.

ELIGIBILITY:
Inclusion Criteria:

* Monthly household income below one half of the median of those in Hong Kong
* Children aged between 5 to 7
* Both children and at least one of their parents agreed to participate in the program

Exclusion Criteria:

* Children or parents with physical disability or mental disorders

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Child Cognitive Development and Behaviour Regulation at 8 weeks | (1) Pretest baseline, and (2) through intervention completion, 8 weeks
  Assessed by counting test and head-shoulder-knee-toe test

SECONDARY OUTCOMES:
Change from Baseline Parental Stress at 8 weeks and at 3 months | (1) Pretest baseline, and (2) 3-month follow up after intervention completion
  Assessed by parent-reported scale, named Parenting Stress Index-Short Form (PSI-SF), assessing the level of parenting stress from different sources of difficulties.
  Total Stress (TS) score and three sub-scores, including Parental Distress (PD), Parental-Child Dysfunctional Interaction (PCDI) and Difficult Child (DC), are reported.
  For the range of TS, the minimum score is 36 and the maximum score is 180. Higher values represent a higher level of total parenting stress.
  For the range of PD, PCDI and DC, the minimum scores are 12 and the maximum scores are 60. Higher values represent a higher level of parenting stress respectively from the source of parental distress, parental-child dysfunctional interaction, and difficult child.
  Three sub-scores are summed to compute a total score.
Change from Baseline Parent Depression at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by parent-reported scale, named Patient Health Questionnaire-9 (PHQ-9), assessing the construct of parent's depression symptoms, directly based on the nine diagnostic criteria for major depressive disorder in the DSM-IV (Diagnostic and Statistical Manual Fourth Edition).
  One total score is reported. For the range of the total score, the minimum score is 0 and the maximum score is 27. Higher values represent parents' more severe level of depression symptoms.
Change from Baseline Mindfulness in Parenting at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by parent-reported scale, named Interpersonal Mindfulness in Parenting (IM-P) scale, assessing the construct of parent's quality of mindfulness specific to his or her family context.
  The total score and four subscale scores, including Compassion for Child (CC), Emotional Awareness in Parenting (EAP), Nonjudgmental Acceptance in Parenting (NAP) and Listening with Full Awareness (LFA), are reported.
  The range of the total score is 23 to 115. Higher values represent parents' better quality of mindfulness in parenting.
  The range of CC is 7 to 35. Higher values represent parents' better quality of compassion for child.
  The range of EAP and NAP is 6 to 30. Higher values respectively represent parents' better quality of emotional awareness in parenting and nonjudgmental acceptance in parenting.
  The range of LFA is 4 to 20. Higher values represent parents' better quality of listening with full awareness.
  Four subscale scores are summed to compute a total score.
Change from Baseline Physiological Stress indicated by salivary cortisol at 8 weeks | (1) Pretest baseline, (2) through intervention completion, 8 weeks
  Assessed by enzyme-linked immunoassay kit
Change from Baseline Physiological Stress indicated by heart rate variability at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by electrocardiogram (ECG)
Change from Baseline Family Functioning at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by parent-reported scale, named Family APGAR scale, assessing parent's satisfaction of family functions.
  One total score is reported. For the range of the total score, the minimum score is 0 and the maximum score is 10.
  Higher values represent parent's better satisfaction of family functions.
Change from Baseline Child Behavior Problem at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by parent-reported scale, named Child Behavior Checklist (CBCL), assessing parents' ratings of their children's behavior problems.
  The Total Problem, and seven subscale scores, including Internalizing Problems, Externalizing Problems, Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Attention Problems, and Aggressive Behavior, are reported.
  For the range of Total Problem and all subscale scores, including Internalizing Problems, Externalizing Problems, Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Attention Problems, and Aggressive Behavior, the minimum scores are 0 and the maximum scores are 1. Higher values respectively represent children's more severe level of overall behavioral problems, Internalizing Problems, Externalizing Problems, Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Attention Problems, and Aggressive Behavior.
  All of them are calculated as the sum of corresponding scale items, and standardized.
Change from Baseline Child Attention at 8 weeks and at 3 months | (1) Pretest baseline, (2) through intervention completion, 8 weeks, and (3) 3-month follow up after intervention completion
  Assessed by computer-aided Attention Network Test (ANT), assessing children's efficiency of attention networks according to their response time to stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Hay-ming Herman Lo, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Corrected according to Advisory Issues (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03662867/Prot_SAP_000.pdf